CLINICAL TRIAL: NCT06227390
Title: Clinical and Radiographic Outcomes of Partial Pulpotomy Procedure in Primary Molars Utilizing Different Capping Materials and Different Restorative Methods: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Outcomes of Partial Pulpotomy Procedure in Primary Molars Utilizing Different Capping Materials and Different Restorative Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Ali Elsharkawy, demonstrator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-005
Record Dates: First submitted 2023-12-22; First posted 2024-01-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-01

CONDITIONS: Pulp Disease, Dental
Keywords: partial pulpotomy
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MTA and stainless-steel crown (Experimental)
  Interventions: Procedure: partial pulpotomy
- Biodentine® and stainless-steel crown (Experimental)
  Interventions: Procedure: partial pulpotomy
- TheraCal PT® and stainless-steel crown (Experimental)
  Interventions: Procedure: partial pulpotomy
- MTA and glass ionomer restoration (Experimental)
  Interventions: Procedure: partial pulpotomy
- Biodentine® and glass ionomer restoration (Experimental)
  Interventions: Procedure: partial pulpotomy
- TheraCal PT® and glass ionomer (Experimental)
  Interventions: Procedure: partial pulpotomy

INTERVENTIONS:
Procedure: partial pulpotomy — 2-3 mm of the coronal pulp tissue is removed leaving healthy vital pulp tissue that is dressed with a dental biomaterial that maintains pulpal vitality and promotes repair

SUMMARY:
the goal of this clinical trial is to compare clinical and radiographic outcomes of partial pulpotomy in vital primary molars using TheraCal PT®, Biodentin® and NeoPUTTY® MTA , followed by glass ionomer restoration only or glass ionomer restoration and stainless-steel crown.

DETAILED DESCRIPTION:
* Primary teeth act as natural space maintainers for the subsequent dentition, they also aid in mastication, satisfactory esthetics and proper articulation of letters. So, it is of prime importance to maintain and preserve their vitality and function through vital pulp therapy (VPT). Ideal VPT materials would sustain pulp vitality, encourage pulp healing. Due to their biocompatibility, bioactivity, and superior sealing capacity, tricalcium silicates (TCSs), such as mineral trioxide aggregate (MTA) and Biodentine®, are currently the most widely used materials for VPT in permanent and primary teeth.Other calcium silicate-based compounds, such as TheraCal PT®, have recently been introduced to the market. TheraCal PT®, a dual-cured variation of its light-cured predecessor Theracal LC®, has improved its chemical capabilities to mitigate the potential harmful consequences of leaving un polymerized monomers.
* The best course of action for primary molars with deep carious lesions that aren't exhibiting any symptoms or indicators of irreversible pulpitis has posed challenges for years. With pulp capping and pulpotomy available as options for primary teeth, and partial pulpotomy in young permanent teeth according to the American Academy of Pediatric Dentistry (AAPD) guidelines for vital pulp therapy. A less invasive version of pulpotomy which is partial pulpotomy uses more conservative theories and biologic principles to produce better clinical results
* New iterations of calcium silicate-based materials have been created for usage as vital pulp therapy material due to their advantageous biological, physical, and mechanical qualities. Additionally, they promote growth factor production and differentiation into odontoblast like cells .
* TheraCal PT® advantages include that it has a hydrophilic matrix which releases Calcium ions. Koutroulis et al.,stated that the increased antibacterial efficacy and calcium release are strongly linked. Also, Calcium release has been linked to the biological characteristics of hydraulic cements because it promotes the differentiation potential of dental pulp cells and enhances mineralization, which results in deposition of a dentine-like barrier on the pulp's surface on the long-term. The other advantage that it increases the pH which provides anti-bacterial activity.
* there is lack of evidence in partial pulpotomy in treatment of carious primary teeth, the materials that could be used in it and necessity of using crown after it.
* this clinical trial will be performed to provide evidence based answer for treatment of primary molars using partial pulpotomy the materials that could be used in it and necessity of using crown after it.

  -• Children will be allocated into either one of the groups of partial pulpotomy depending on the medicament used as follows:
  * Group 1A: (control group) MTA and stainless-steel crown.
  * Group 1B: MTA and glass ionomer restoration.
  * Group 2A: Biodentin® and stainless-steel crown.
  * Group 2B: Biodentin® and glass ionomer restoration.
  * Group 3A: TheraCal PT® and stainless-steel crown.
  * Group 3B: TheraCal PT® and glass ionomer restoration. All of the medicaments will be applied according to the manufacturer's instructions and gently placed over the pulp tissue to a thickness of 2mm then the rest of the pulp chamber will be filled with glass ionomer cement
* Clinical follow up after 3,6,9 and12 months while radiographic follow up every 6 months.

  * Parents will be asked if any complains occurred between follow up visits by phone

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients aged 4-7-years old.
2. Cooperative patients (Frankle scale + and ++)
3. Asymptomatic primary molar with deep caries requiring vital pulp therapy

Exclusion Criteria:

* presence of any of the following:

  1. History of spontaneous lingering pain, swelling, or sinus tract.
  2. Pathological mobility.
  3. pain on percussion.
  4. Furcation or periapical radiolucency.
  5. pathological root resorption

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate and Compare clinical outcomes of TheraCal PT®, Biodentin® and NeoPUTTY®, followed by glass ionomer restoration only or glass ionomer restoration and stainless-steel crown.in partial pulpotomy in vital primary molars | 1 year
  method of measurement: presence or absence of pain, swelling, fistula, mobility unit of measurement: yes or no

SECONDARY OUTCOMES:
Evaluate and compare Radiographic outcomes of TheraCal PT®, Biodentin® and NeoPUTTY® MTA, followed by glass ionomer restoration only or glass ionomer restoration and stainless-steel crown in partial pulpotomy in vital primary molars | 1year
  method of measurement: comparing pre and post operative radiographs unit of measurement: presence of furcation or periapical radiolucency, pathologic external root resorption, or internal resorption

CONTACTS AND LOCATIONS:
Locations (1):
- the British University in Egypt, Cairo, Egypt